CLINICAL TRIAL: NCT05265013
Title: A Phase 2 Single-arm Study of ASP-1929 Photoimmunotherapy Combined With Pembrolizumab in Patients With Locoregional Recurrent Squamous Cell Carcinoma of the Head and Neck, With or Without Metastases, Not Amenable to Curative Local Treatment
Brief Title: ASP-1929 Photoimmunotherapy Combined With Pembrolizumab in Patients With Recurrent Head and Neck Cancer, With or Without Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Rakuten Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASP-1929-218
Record Dates: First submitted 2022-01-25; First posted 2022-03-03 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
Keywords: Rakuten Medical; ASP-1929; PIT; Photoimmunotherapy; HNC; HNSCC; Head and neck; pembrolizumab
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: ASP-1929 Photoimmunotherapy Combined With Pembrolizumab
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ASP-1929 Photoimmunotherapy Combined With Pembrolizumab (Experimental): Patients will receive the approved label dose of pembrolizumab, which is administered every 3 weeks on days 1 and 22 of each treatment cycle.
  On Day 8 of each cycle, patients will receive ASP-1929 followed by illumination at accessible tumor sites using the investigational PIT690 Laser System on Day 9.
  Each treatment cycle, which is driven by ASP-1929 PIT frequency of administration, will last 42 days. Patients will be treated with ASP-1929 PIT and pembrolizumab for up to 12 months with a maximum of 8 treatment cycles.
  Interventions: Combination Product: ASP-1929 Photoimmunotherapy; Biological: pembrolizumab

INTERVENTIONS:
Combination Product: ASP-1929 Photoimmunotherapy — ASP-1929 640 mg/m^2 IV infusion followed by illumination with light dose of 50 J/cm^2 for superficial lesions and 100 J/cm for interstitial lesions within 24 +/- 4 hours after the end of ASP-1929 infusion
  Other Names: cetuximab sarotalocan, PIT690 Laser System
Biological: pembrolizumab — 200 mg every three weeks on days 1 and 22 of each 6-week cycle, 30 minute IV infusion
  Other Names: Keytruda

SUMMARY:
A Phase 2 Single-arm Study of ASP-1929 Photoimmunotherapy Combined With Pembrolizumab in Patients With Locoregional Recurrent Squamous Cell Carcinoma of the Head and Neck, With or Without Metastases, Not Amenable to Curative Local Treatment

DETAILED DESCRIPTION:
A Single-arm Study of ASP-1929 Photoimmunotherapy Combined With Pembrolizumab.

Patients will receive the approved label dose of pembrolizumab, which is administered every 3 weeks on days 1 and 22 of each treatment cycle.

On Day 8 of each cycle, patients will receive ASP-1929 followed by illumination at accessible tumor sites using the investigational PIT690 Laser System on Day 9.

Each treatment cycle, which is driven by ASP-1929 PIT frequency of administration, will last 42 days. Patients will be treated with ASP-1929 PIT and pembrolizumab for up to 12 months with a maximum of 8 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Male or female ≥ 20 years of age at the time of signing informed consent.
3. Have histologically or cytologically confirmed and diagnosed locoregional recurrent or second primary squamous cell carcinoma of the head and neck, not amenable to curative local treatment (ie, surgery and radiation therapy) per treatment guidelines. Patients with distant metastases are eligible.
4. Have provided tissue for biomarker analysis from a fresh core or excisional biopsy. A newly obtained screening biopsy (prior to start of study treatment with no intervening anticancer treatment from time of biopsy collection to C1D1) is strongly preferred but an archival sample is acceptable provided it has been collected within ≤ 6 months of enrollment and no intervening anticancer treatment has occurred within that timeframe or upon agreement from the Sponsor.
5. Disease progression after treatment with a platinum-containing regimen for recurrent (disease not amenable to curative treatment)/metastatic disease. Note: disease progression may occur at any time during or after a platinum-containing regimen (eg, carboplatin or cisplatin) which was administered in the recurrent/metastatic setting.

   Note: Patients who were ineligible or unable to receive platinum therapy may be eligible after failing or progressing after suitable alternative systemic therapy (eg, 5-FU, cetuximab).
6. Anti-PD-1 treatment naive.
7. Completed prior curative radiation therapy for treatment of the head and neck region, unless, in the opinion of the investigator, the use of radiation therapy was contraindicated or not recommended.
8. At least one recurrent head and neck tumor that is both accessible for illumination (as assessed by investigator) and radiographically measurable by RECIST v1.1 as assessed by an independent central reviewer (ICR) and the investigator. Lesions located in a previously irradiated area are considered measurable if progression has been demonstrated.

   1. Accessible tumors may be superficial lesions that are amenable to superficial illumination, regional metastatic lesions such as accessible lymph nodes, or deeper tumors that may be illuminated interstitially using cylindrical diffusers.
   2. Tumors that require needle catheters to go through bone (except tumors inside paranasal sinuses), arteries, major veins, eye globes, dura, or brain (including perineural invasion extending to the skull base) are not suitable for PIT illumination.
9. Combined positive score (CPS) ≥ 1 (as determined by a Taiwan Food and Drug Administration/TFDA approved test).
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at the time of screening.
11. Life expectancy ≥ 3 months based on investigator judgement.
12. Adequate organ function laboratory values as described below (all screening labs should be performed ≤ 7 days of C1D1):

    1. Hematology: Adequate bone marrow function as shown by absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, hemoglobin (Hb) ≥ 9 g/dL. Transfusions and growth factors must not be used within 2 weeks prior to C1D1 to meet these requirements.
    2. Hepatic: Alkaline phosphatase (ALP) ≤ 2 times upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (≤ 5 times ULN for patients with liver metastases), and total serum bilirubin ≤ 2 mg/dL (unless the patient has Gilbert's disease).
    3. Renal: estimated glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m² to be calculated per the CKD-EPI equation below:

       GFR = 141 * min (Scr/κ,1)ᵅ * max(Scr/κ, 1)-¹.²⁰⁹ * 0.993ᵃᵍᵉ * 1.018 [if female] * 1.159 [if Black] Note: Scr is serum creatinine (mg/dL), κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1.
    4. Coagulation: International Normalized Ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN, unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants.
13. Female patients of childbearing potential must not be pregnant (confirmed by negative pregnancy test [urine or serum] at screening) or breastfeeding and must be willing to use 2 methods of highly effective birth control or practice abstinence throughout the study and for 120 days after the last dose of study medication. Females of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
14. Male patients must be sterile or agree to use an adequate method of contraception or practice abstinence starting with the first dose of study medication through 120 days after the last dose of study treatment.

Exclusion Criteria:

Patients will be excluded if any of the following criteria apply:

Medical History

1. Diagnosed and/or treated for an additional malignancy within 5 years prior to study C1D1, except for those with a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ). Patients with a history of other prior cancer with no evidence of disease may be eligible based on discussion with the medical monitor.
2. Tumor invading a major blood vessel unless the vessel has been embolized or surgically ligated to prevent hemorrhage; must not have involvement of the common or internal carotid arteries defined as invasion, encasement, or direct contact (lack of a radiographically visible plane between the tumor and carotid artery). Decision to exclude may be determined either by a central reviewer or by the investigator.
3. Tumors inappropriate for ASP-1929 PIT treatment, including those in the brain or dura, with perineural involvement at the skull base, CNS (Central nervous system) disease, or disease in the orbit (if the eye has been previously removed, consult with the medical monitor before excluding). Decision to exclude may be determined by a central reviewer or the investigator.
4. Known or active central nervous system metastases and/or carcinomatous meningitis.
5. Active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.

   Note: Patients with type I diabetes mellitus or hypothyroidism requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are not excluded.
6. Evidence of interstitial lung disease or current active, non-infectious pneumonitis.
7. Active infection requiring systemic therapies such as antibiotic, antifungal, or antiviral intervention which in the opinion of the Investigator precludes the patient from participating in the clinical trial.
8. Prior allogeneic tissue/solid organ transplant.
9. History of significant (≥ grade 3) infusion reactions to anti-EGFR (EGFR, epidermal growth factor receptor) antibodies.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ASP-1929 or pembrolizumab.
11. Known history of testing positive for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
12. Known infection or detection of active Hepatitis B (eg, HBsAg positive), active Hepatitis C (eg, RNA [qualitative]), or SARS-CoV-2 (qualitative).
13. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Any other condition which, in the investigator's opinion, deems the patient an unsuitable candidate to receive pembrolizumab, ASP-1929, and/or be exposed to illumination, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.

    Prior and Concomitant Procedures
15. Major surgery or significant traumatic injury within 4 weeks prior to C1D1, or anticipation of the need for major surgery during the study.

    Note: If patient has had major surgery, they must have recovered adequately (as determined by the investigator) from the toxicity and/or complications before C1D1.
16. Requiring future examinations or treatments within 4 weeks after an ASP-1929 PIT treatment cycle exposing the patient to high intensity light (eg, eye examinations, surgical procedures that are unrelated to the ASP-1929 PIT treatment, the disease under study, or the study overall).

    Prior and Concomitant Medications
17. Prior receipt of anticancer treatment as follows:

    1. Prior systemic chemotherapy or targeted small molecule therapy or radiation therapy within 2 weeks of C1D1 or has not recovered (ie, ≤ Grade 1 or at baseline) from adverse events due to previously administered agent.
    2. Prior anticancer monoclonal antibody therapy or investigational agent or intervention within 4 weeks of C1D1 or has not recovered (ie, ≤ Grade 1 or at baseline) from adverse events due to previously administered agent.
    3. Prior receipt of ASP-1929 at any time.
18. Receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to C1D1.
19. Received a live, attenuated vaccine within 4 weeks before C1D1 or anticipation of receiving a live, attenuated vaccine during the study (based on known medical history).

    Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (eg, Flu-Mist®) are live attenuated vaccines and are not allowed.
20. Unwilling or unable to follow protocol requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR-PIT) | 24 months
  the proportion of patients with confirmed PIT-treated tumor response of complete response (CR) or partial response (PR) per RECIST 1.1, as assessed by central reviewer.

SECONDARY OUTCOMES:
Duration of Response, for PIT-treated lesions | 24 months
  Duration of Response (DoR; Duration of Response is defined as the time from first response (CR or PR) to the time of disease progression (PD) of PIT-treated lesions per RECIST 1.1, as assessed by central reviewer.
Assess effects on tumor response, for PIT-treated lesions | 24 months
  Disease Control Rate (complete response, CR + partial response, PR + stable disease, SD) for PIT-treated lesions per RECIST 1.1, as assessed by central reviewer.
Assess effects on tumor response, Confirmed ORR for all lesions | 24 months
  For all lesions per RECIST 1.1, as assessed by central reviewer:
  • Confirmed ORR (CR or PR)
Assess effects on tumor response, Disease control rate for all lesions | 24 months
  For all lesions per RECIST 1.1, as assessed by central reviewer:
  • Disease control rate (DCR)
Assess effects on tumor response, DoR for all lesions | 24 months
  For all lesions per RECIST 1.1, as assessed by central reviewer:
  • DoR
Assess effects on survival, PFS | 24 months
  Progression-free Survival (PFS)
Assess effects on survival, OS | 24 months
  Overall Survival (OS)
Characterize safety and tolerability | 24 months
  Proportion of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), serious adverse events (SAEs) by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Assess effects on quality of life, European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | 12 months
  Change from baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). It has four-point scales for the first 28 items. The minimum value is 1 and maximum value is 4. Higher scores mean a worse outcome. Overall health was evaluated as a 7-point response scale as the other two questions in that scale. The minimum value is 1 and maximum value is 7. Higher scores mean a better outcome.
Assess effects on quality of life, EORTC head and neck specific module (EORTC QLQ H&N 35) | 12 months
  Change from baseline in EORTC head and neck specific module (EORTC QLQ H&N 35). It has 4-point scales for the first 30 items. The minimum value is 1 and maximum value is 4. It has 2-point scales for the last 5 items. The minimum value is 1 and maximum value is 2. For all items and scales, high scores indicate more problems.
Assess effects on quality of life, Functional Assessment of Cancer Therapy Head & Neck Cancer Symptom Index - 10 Item (FHNSI-10) | 12 months
  Proportion of patients who achieve a clinically meaningful benefit in symptoms, as measured by a 5-point improvement in Functional Assessment of Cancer Therapy Head & Neck Cancer Symptom Index - 10 Item (FHNSI-10) from baseline to measured best assessment. The minimum value is 0 and maximum value is 4. Higher scores mean a worse outcome.
Characterize population pharmacokinetics of ASP-1929, AUC₀-ₜ (AUC, area under the concentration-time curve) | 12 months
  Area under the concentration-time curve from time 0 through the last measurable time point.
Characterize population pharmacokinetics of ASP-1929, AUC₀-₂₆ | 12 months
  Area under the concentration-time curve from time 0 until 26 hours after infusion initiation (just prior to light treatment).
Characterize population pharmacokinetics of ASP-1929, AUC₀-∞ | 12 months
  Area under the concentration-time curve from time 0 through the last measurable time point and extrapolated to infinity.
Characterize population pharmacokinetics of ASP-1929, AUCₐₗₗ | 12 months
  Area under the concentration-time curve using all available data from 0 through 2 weeks post dose.
Characterize population pharmacokinetics of ASP-1929, Cₘₐₓ (maximum observed drug concentration) | 12 months
  Maximum observed concentration.
Characterize population pharmacokinetics of ASP-1929, tₘₐₓ (time to maximal concentration) | 12 months
  Time of maximum observed concentration.
Characterize population pharmacokinetics of ASP-1929, t₁/₂ (mean terminal elimination half-life) | 12 months
  The observed terminal elimination half-life.
Characterize population pharmacokinetics of ASP-1929, CL (volume of serum cleared of drug per unit time) | 12 months
  The volume of serum cleared of drug per unit time following IV dosing (ASP-1929 only).
Characterize population pharmacokinetics of ASP-1929, Vₛₛ (volume of distribution at steady state following intravenous administration) | 12 months
  Volume of distribution following IV dosing (ASP-1929 only).
Characterize presence of anti-drug antibodies (ADA) | 24 months
  Proportion of patients with anti-ASP-1929 antibodies.

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No